CLINICAL TRIAL: NCT03979586
Title: Intradermal Delivery of Fractional CO2 Laser-assisted Hyaluronic Acid in Facial Skin Remodeling
Brief Title: Laser-assisted Hyaluronic Acid Delivery by Fractional CO2 Laser in Facial Skin Remodeling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-17; RC12_0036 (Registry Identifier: APHM)
Record Dates: First submitted 2019-05-02; First posted 2019-06-07 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Facial Skin Remodeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient phototype I to IV (Experimental): The study will be conducted in the Laser Dermatological and Plastic Center of the Conception Hospital in Marseille. It will be a prospective, controlled, hemiface, single-blind, independent-evaluator pilot study of 20 patients, 30 to 70 years old, with phototype I to IV (Fitzpatrick scale). By this study in hemiface, each patient will be his own witness. Neither the patient nor the examining doctor will know the choice of the hemiface of application of hyaluronic acid. This will be a single-blind study with independent evaluator. Patients will be included for 3 months, and followed for a period of 3 months.
  Interventions: Other: Laser-assisted hyaluronic acid delivery

INTERVENTIONS:
Other: Laser-assisted hyaluronic acid delivery — The facial skin remodeling corresponds to a request for repair treatment on the stigmas of heliodermia, irregularity of cutaneous texture, dyschromias, loss of radiance of the complexion, fine lines, as well as on the fine scars of the face for example, the finely depressed cicatrices sequellaires acne.

SUMMARY:
The main endpoint will be to evaluate the efficacy of laser-assisted hyaluronic acid delivery by fractional CO2 laser in facial skin remodeling. The secondary endpoint will be to confirm the safety of this protocol compared to a standard treatment by fractional CO2 laser.

DETAILED DESCRIPTION:
Fractional CO2 lasers are already used in skin remodeling. They can also create vertical channels to enhance topical drug delivery deep into the dermis. Combining the efficacy of fractional CO2 laser to laser-assisted hyaluronic acid delivery has not yet being studied, the combination of these two techniques could improve facial skin remodeling.

The main endpoint will be to evaluate the efficacy of laser-assisted hyaluronic acid delivery by fractional CO2 laser in facial skin remodeling. The secondary endpoint will be to confirm the safety of this protocol compared to a standard treatment by fractional CO2 laser.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Laser Center for facial skin remodeling,
* aged from 30 to 70 years old,
* with phototype I to IV (Fitzpatrick scale),
* agreeing to participate in this study, signing the informed consent form
* not fitting in any non-inclusion criterion

Exclusion Criteria:

* Pregnancy or breastfeeding,
* active infection, history of oral or genital herpes
* suspected neoplasia,
* active inflammatory or infectious facial dermatitis,
* oral retinoid treatment in the last 6 months,
* phototype V or VI (Fitzpatrick scale)
* age <30 years or> 70 years,
* patients under guardianship or curatorship,
* hemostasis disorders, thrombolytic or anticoagulant therapy, c
* ongenital methaemoglobinaemia,
* porphyria,
* known hypersensitivity to hyaluronic acid, local anesthetics of the amide group or to any other component of Anesderm cream Ge 5%

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Measurement of the improvment of one of the skin remodeling parameters (cutaneous texture, firmness, fine lines, radiance) using a scale from 0 to 10 | 3 months
  The primary judgment criterion will be the improvement at 3 months of at least one of the skin remodeling parameters (cutaneous texture, firmness, fine lines, radiance) at least 2 points greater (on a scale of 0 to 10) on fractional laser and hyaluronic acid-treated hemiface compared to fractional laser and control saline-treated hemiface.

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France